CLINICAL TRIAL: NCT00276978
Title: Aripiprazole Augmentation Therapy in Treatment-resistant Depression
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Initiation of study was stopped due to administrative reasons before first subject was enrolled.
Sponsor: University Hospital Freiburg (Other)
Responsible Party: Principal Investigator, Claus Normann, Prof. Dr., University Hospital Freiburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Aripiprazole Augmentation
Record Dates: First submitted 2006-01-11; First posted 2006-01-13 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Therapy-resistant Depression
Keywords: Therapy-resistant Depression; add-on therapy depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): Aripiprazol augmentation therapy
  Interventions: Drug: Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole — Addition of Aripiprazole 10 mg to concurrent medication
  Other Names: Abilify

SUMMARY:
20 therapy-refractory patients with major depression will be treated for 3 weeks with Aripiprazole 10 mg/d. Effectivity will be assessed using a pre-post comparison of different psychopathological rating scales and patient adherence.

DETAILED DESCRIPTION:
This will be an open pilot study using pre-post comparison. 20 treatment-refractory patients with major depression diagnosed by DSM-IV will be included. Psychotic features of depression will be excluded by a score of 2 or less in the PANSS subscales P1, P3 and P6. Treatment resistance as defined by history of non-response to two antidepressants from different classes at an acceptable dose and period is confirmed retrospectively. If possible, treatment compliance should be confirmed by plasma level examination. After informed consent, visit 1 is performed on day 0 (inclusion criteria, history, demographics, physical examination, vital signs, HAMD, MADRS, CGI, BDI, lab). Study medication is started on day 1, the antidepressive therapy is continued at stable dose until the end of the study. Patients will receive an adjunctive augmentation therapy of 10 mg/d aripiprazole. Study visits will be performed on days 3, 7, 14 and 21 (visits 2-5: vital signs, HAMD, MADRS, CGI, BDI, lab). In addition to the HAM-D and MADRS scores, patients will perform a self-rating (BDI). Aripiprazole plasma levels will be measured at the end of the treatment period to assess compliance and to detect a putative correlation between drug plasma levels and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* major depression without psychotic features (DSM-IV definition)
* therapy resistance (two courses of antidepressants from different classes for more than 3 weeks in adequate dose)
* HAM-D score greater/equal than 17
* age 18-70

Exclusion Criteria:

* bipolar disorder
* active alcohol or illicit drug use
* female without effective contraception
* severe medical conditions
* psychotic features

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2009-11 (Estimated); Study Completion 2009-11 (Estimated)

PRIMARY OUTCOMES:
rate of response as defined by a more or equal 50 % reduction of baseline HAM-D (Hamilton Depression Rating scale) | 4 wks

CONTACTS AND LOCATIONS:
Overall Officials: Claus Normann, MD, Principal Investigator — Department of Psychiatry, University of Freiburg
Locations (1):
- Dept. of Psychiatry, University of Freiburg, Freiburg im Breisgau, Germany